CLINICAL TRIAL: NCT02777775
Title: Targeting the Mechanisms Underlying Cutaneous Neurofibroma Formation in NF1: A Clinical Translational Approach.
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Matthew Steensma, Dr. Matthew Steensma, Corewell Health West
Other Study IDs: 2014-295
Record Dates: First submitted 2015-01-21; First posted 2016-05-19 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous Neurofibromas; Neurofibromatosis Type 1; Plexiform Neurofibromas
Keywords: NF1; CNF; PNF; Skin Tumors
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Harvesting CNFs from 3 groups of subjects in order to obtain a minimum of 18 tumors in three size categories: <5mm, 5-10mm, and >1cm
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Skin Biopsy — The procedure to sample the cutaneous neurofibroma involves a skin incision and will take approximately 10 to 15 minutes. The tissue will be taken in the following way:
  * The skin area will be cleaned
  * The skin area will be numbed (by either a numbing cream or a tiny numbing shot)
  * Cutaneous (skin) Neurofibroma: will be taken via a small incision and removal of the neurofibroma whenever possible.
  * A small piece of normal (skin) tissue will be numbed as above and taken using a special skin biopsy device.
  Afterward, the area will be cleaned and the skin put back together with medical super glue or 1 to 2 dissolvable stitches that will dissolve as the incision heals, they do not require removal. The purpose of taking this piece of skin is to compare normal skin with the skin of a cutaneous neurofibroma.

SUMMARY:
The purpose of the research study is intended to use specimens (such as tissue) and medical information in the Laboratory of Musculoskeletal Oncology at the Van Andel Research Institute for laboratory research in Grand Rapids, Michigan. Small tissue samples of cutaneous neurofibromas will be collected as part of this research. The samples will help researchers learn more about cutaneous neurofibroma and help them better understand NF1. There are many different types of studies, both now and in the future, that can be done using the specimens the investigators receive. These include using the specimens and information to look for new ways to diagnose and treat Neurofibromatosis Type 1 (NF1). The specimens may be used to study how genes affect health and disease, or how genes affect the way a disease or condition responds to treatment. Some of these studies may lead to new products, such as treatments or tests for diseases. Through this study, the investigators hope to find better ways to understand and treat NF1 in the future.

DETAILED DESCRIPTION:
Skin tumors in Neurofibromatosis Type 1 (NF1) are very common and diminish quality of life. Apart from surgery, very few treatment options exist. In comparison to other types of tumors in NF1, skin tumors receive less attention in the research world because they almost never turn into cancer. Under the microscope, skin tumors and plexiform tumors look similar, however they do not share the same growth potential, nor do they appear at the same time during development. These differences suggest that skin tumors are driven by different factors than plexiform tumors.

In this study the investigators will be harvesting CNFs from 3 groups of subjects in order to obtain a minimum of 18 tumors in three size categories: <5mm, 5-10mm, and >1cm. These sizes were selected based on the variable natural history of CNF progression where incipient lesions (typically <5mm) are more numerous and demonstrate a less aggressive growth pattern, whereas the intermediate group (5-10mm) represent a transition state towards growth to larger (>1cm) lesions. Interestingly, CNF growth tends to stall out at 3cm. The investigators plan to do experiments that identify which factors are important to CNF progression, and then find matching drugs that can shrink the tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Any subject with an established diagnosis NF1 and CNFs. The diagnosis may be based on clinical criteria or genetic testing.
2. Age >18 years.

Exclusion Criteria:

1. Adults with diminished decision-making capacity with no defined legal guardian.
2. Prisoners.
3. Pregnant women.

3) Breastfeeding mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone with an established diagnosis NF1 and CNFs. The diagnosis may be based on clinical criteria or genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-05; Primary Completion 2025-06 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
Tissue Harvesting via Tissue Excision - up to 74 CNFs will be collected from patients to obtain 8 tumors in three size categories: <5mm, 5-10mm, and >1cm. CNFs will be determined based on examiner's experience. | 2 Years
  Identify which genomic factors are important to CNF progression, and find matching drugs that can shrink the tumors and improve quality of life.

SECONDARY OUTCOMES:
UV Exposure and NF1 History Questionaires | 2 Years
  Measuring the relationship between sun exposure and CNF growth and development.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Steensma, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospital Group, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No